CLINICAL TRIAL: NCT03221062
Title: Comparison of the Pathological Stage and Clinical Outcome of en Bloc Transurethral Resection by HybridKnife or Laser Versus Conventional Transurethral Resection for NMIBC: a Prospective, Single Centre, Randomized Study
Brief Title: "En Bloc" Resection of NMIBC: a Prospective， Single Centre，Randomized Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jia Hu, Principal Investigator, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JHu
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser en Bloc Resection (Experimental): Laser en Bloc Resection of bladder tumor(laser ERBT)
  Interventions: Device: Laser en Bloc Resection
- Hydroknife en Bloc Resection (Experimental): Hydroknife en Bloc Resection of bladder tumor (Hydroknife ERBT)
  Interventions: Device: Laser en Bloc Resection
- conventional transurethral resection (Experimental): conventional transurethral resection of bladder tumor(cTURBT)
  Interventions: Device: Laser en Bloc Resection

INTERVENTIONS:
Device: Laser en Bloc Resection — Procedure: Laser en Bloc Resection of bladder tumor Procedure: Hydroknife transurethral resection of bladder tumor Procedure: conventional transurethral resection
  Other Names: Hydroknife en Bloc Resection; conventional transurethral resection

SUMMARY:
The traditional method of choice for intravesical resection of bladder tumors is conventional transurethral resection of bladder tumor (cTURBT). However, there has long been an ambition to overcome its biggest limitation, tumor fragmentation. Possible consequences include cell seeding and poor specimen quality, including missing detrusor muscle, thermal tissue damage, and tissue fragmentation. En bloc resection of bladder tumor (ERBT) represents an alternative technique for resection of bladder tumors. There is no doubt that ERBT has huge potential. ERBT provides specimens of high quality that are easy for pathologists to read. In theory, this may sustainably change the view on secondary resection, lead to faster decisions on subsequent treatments, and influence patient prognosis. Thus, there is an urgent need to compare ERBT with cTURBT in a thoroughly planned trial.

DETAILED DESCRIPTION:
Urothelial bladder cancer (UBC) represents a major worldwide healthcare challenge in western countries as well as in developing countries, both oncologically and economically. Initially, most patients present with nonmuscle invasive bladder cancer (NMIBC) with disease confined to the mucosa (stage Ta, carcinoma in situ) or submucosa (T1) characterized by a far lower mortality rate compared with muscle invasive bladder cancer (MIBC).The vast majority of newly diagnosed are non-muscle bladder cancers (NMIBC) which represents about 75% and can be treated with transurethral resection of bladder tumors (TURBT). Therefore, correct initial staging is critical. The quality of TURBT strongly determines patient prognosis and overall treatment.

Conventional transurethral resection of bladder tumors (cTURBT) causes fragmentation. Possible consequences include cell seeding and poor specimen quality, including missing detrusor muscle, thermal tissue damage, and tissue fragmentation. ERBT is developing concept as an alternative to conventional TURBT. En bloc is identified by using various energy sources or modified resection loops as a promising technique. Such as HybridKnife or laser.

The question has been raised as to whether ERBT is ready for guideline implementation. Only two prospective, randomized trials on ERBT have been published. However, there are details on statistical preparation, patient selection, and definitions of primary and secondry goals are missing. Thus, there is still an urgent need to compare ERBT with cTURBT in a thoroughly planned trial.

This study will be conducted in a single centre at Department of Urology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China.

Eligible patient presented with papillary bladder tumor will be asked to participate in this study and will be provided with an informed consent form in line with Good Clinical Practise and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological or histological diagnosis by cystoscopy of primary non-muscle invasive bladder urothelial carcinoma (Ta, T1);
2. Imaging examinations showed the bladder muscle has not been affected, no lymph node metastasis or distant metastasis;
3. Diameter of tumor 1-3cm
4. Number of lesions≤3 (The position of small lesions relatively concentrated as one place)
5. Patients who agree to ERBT or cTURBT surgery, and will be effected to the postoperative follow-up treatment such as conventional infusion after the operation

Exclusion Criteria:

1. Tis or non-transitional epithelial tumors
2. Pathological or imaging examinations showed the bladder muscle has not been affected
3. There has surgery contraindications, such as bladder fibrosis
4. Diameter of tumor >3cm or <1cm
5. Number of lesions>3
6. Anteriorly located tumor
7. Received chemotherapy or BCG perfusion therapy in the nearly 3 months
8. Poor performance status is difficult to tolerate surgery
9. The patient refused to sign a consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
The pathological staging assessment | one week
  The pathological staging assessment for ERBT or cTURBT procedure
The recurrence rate assessment at resection sites | two year
  The recurrence rate assessment at resection sites for ERBT or cTURBT procedure

SECONDARY OUTCOMES:
periprocedure complications | 2 days
  Modified Clavien scale will be used for reporting and comparison of periprocedure complications(obturator nerve reflection;bladder perforation)

IPD SHARING:
Plan to Share IPD: Undecided